CLINICAL TRIAL: NCT01155154
Title: Antibiotic Prophylaxis for Prevention of Infection in Emergency Department Patients With Simple Hand Lacerations
Brief Title: Antibiotic Prophylaxis for Simple Hand Lacerations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: Staten Island University Hospital (Other); Kings County Hospital Center (Other)
Responsible Party: Principal Investigator, Shahriar Zehtabchi, Professor of Emergency Medicine, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-130
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Simple Hand Lacerations
Keywords: wounds and lacerations; hand; infection; Antibiotics; antibacterial agents
MeSH Terms: conditions — Wounds and Injuries; Lacerations; Infections | interventions — Cephalexin; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- clindamycin (Active Comparator): clindamycin 300 mg (two 150 mg capsules) every 6 hours for 7 days
  Interventions: Drug: clindamycin
- cepahlexin (Active Comparator)
  Interventions: Drug: cephalexin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cephalexin — 500 mg (two 250 mg capsules) every 6 hours for 7 days
  Arms: cepahlexin
Drug: clindamycin — 300 mg of clindamycin (two 150 mg capsules) every 6 hours for 7 days
  Arms: clindamycin
Drug: placebo — Two placebo capsules every 6 hours for 7 days
  Arms: Placebo

SUMMARY:
Research Question: In emergency department patients with simple hand cuts, do prophylactic antibiotics reduce the risk of wound infections?

DETAILED DESCRIPTION:
Simple hand lacerations, defined as hand lacerations that do not involve special structures such as bones, tendons, vessels, or nerves, are common in the emergency departments. The exact rate of infection in such wounds is unclear. It is also not clear whether prescribing prophylactic antibiotics reduces the risk of infection in simple hand lacerations. The objective of this randomized double blind controlled study is to: 1. Identify the rate of infection in simple hand lacerations, 2. Identify factors or wound characteristics that increase the risk of infection, and 3. Assess whether prescribing prophylactic antibiotics decreases the risk of infections in such wounds compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years of age) presenting to the ED with simple hand lacerations. Anatomically, lacerations distal to the radial carpal ligament will be considered "hand" lacerations. "Simple" or "uncomplicated" laceration refers to one that does not involve any special tissue (bone, tendon, blood vessel, or nerve).

Exclusion Criteria:

* Immunocompromised patients (cancer, chemotherapy, transplant, HIV/AIDs)
* Current or recent (within two weeks) use of any antibiotics
* Allergy to clindamycin or cephalexin
* Bites (e.g. dog, cat, or human)
* Lacerations resulted from crush injury
* Lacerations involving bone, tendon, blood vessel, or nerve
* Lacerations inflicted more than 12 hours prior to ED visit
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: shahriar zehtabchi, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (3):
- United States (3):
  - Kings County Hospital Center, Brooklyn, New York
  - State University of New York, Downstate Medical Center, Brooklyn, New York
  - Staten Island University Hospital, Staten Island, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clindamycin | Cepahlexin | Placebo
Started | 25 | 24 | 24
Completed | 25 | 24 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The median age of the subjects was 40 years (quartiles: 29, 53), and 71% were male (n=52).
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin | Cepahlexin | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 24 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [26 to 56] | 42 [32 to 58] | 40 [29 to 52] | 41 [29 to 55.5]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 20 | 63
  >=65 years | 2 | 4 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 5 | 21
  Male | 15 | 18 | 19 | 52
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Wound Infection
Description: Hand lacerations will be examined 10-14 days after initial wound closure and will be assessed for presence of infection.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Clindamycin | Cepahlexin | Placebo
Number analyzed (Participants) | 25 | 24 | 24
participants | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Clindamycin | Cepahlexin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/25 | 1/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin (N=25) | Cepahlexin (N=24) | Placebo (N=24)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
palpitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Metal After-taste in th mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No